CLINICAL TRIAL: NCT05061537
Title: A PHASE 1, OPEN-LABEL, DOSE ESCALATION AND EXPANSION STUDY EVALUATING THE SAFETY AND PHARMACODYNAMICS OF PF-07263689, EITHER ALONE OR IN COMBINATION WITH AN ANTI-PD-1 ANTIBODY, IN PREVIOUSLY TREATED PARTICIPANTS WITH SELECTED LOCALLY ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: Study of PF-07263689 in Participants With Selected Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor due to business decision and not due to any safety concerns with PF-07263689. There are no changes to the risk-benefit for participants who have received PF-07263689 in the study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4651001; OBIR-2 (Other: Alias Study Number)
Record Dates: First submitted 2021-09-22; First posted 2021-09-29 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Renal Cell Cancer; Melanoma; Non-Small-Cell Lung Cancer; Hepatocellular Cancer; Bladder Cancer; Sarcoma; Head and Neck Cancer; Colorectal Cancer; Ovarian Cancer; Squamous Cell Carcinoma
Keywords: Advanced malignancies
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma; Carcinoma, Non-Small-Cell Lung; Liver Neoplasms; Urinary Bladder Neoplasms; Sarcoma; Head and Neck Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Monotherapy dose escalation (Part 1A) (Experimental): Participants will receive PF-07263689 once a week for 4 doses
  Interventions: Biological: PF-07263689
- Combination dose escalation (Part 1B) (Experimental): Participants will receive PF-07263689 intravenous (IV) once week for 4 doses in combination with sasanlimab subcutaneous (SC) once every 4 weeks
  Interventions: Biological: PF-07263689; Biological: Sasanlimab
- Dose expansion (Part 2) - Tumor specific Arm A (Experimental): Participants will receive PF-07263689 IV once week for 4 doses in combination with sasanlimab SC once every 4 weeks
  Interventions: Biological: PF-07263689; Biological: Sasanlimab
- Dose expansion (Part 2) - Tumor specific Arm B (Experimental): Participants will receive PF-07263689 IV once week for 4 doses in combination with sasanlimab SC once every 4 weeks
  Interventions: Biological: PF-07263689; Biological: Sasanlimab
- Dose expansion (Part 2) - Tumor specific Arm C (Experimental): Participants will receive PF-07263689 IV once week for 4 doses in combination with sasanlimab SC once every 4 weeks
  Interventions: Biological: PF-07263689; Biological: Sasanlimab

INTERVENTIONS:
Biological: PF-07263689 — Genetically engineered oncolytic vaccinia virus
Biological: Sasanlimab — A monoclonal antibody that blocks the interaction between PD-1 and PD-L1/ PD-L2
  Arms: Combination dose escalation (Part 1B); Dose expansion (Part 2) - Tumor specific Arm A; Dose expansion (Part 2) - Tumor specific Arm B; Dose expansion (Part 2) - Tumor specific Arm C

SUMMARY:
This is a first-in-human, Phase 1, open label, multicenter, multiple dose, dose escalation and expansion study intended to evaluate the safety, viral load kinetics and shedding, pharmacodynamic, and anti-tumor activity of PF-07263689, either alone or in combination with sasanlimab (an investigational anti-programmed cell death protein 1 [PD-1] antibody), in patients with selected locally advanced or metastatic solid tumors who have exhausted all available standard of care therapies available to them.

The study consists of 2 parts: Part 1 dose escalation for PF-07263689 monotherapy (Part 1A) and in combination with sasanlimab (Part 1B), followed by Part 2 dose expansion for the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of locally advanced or metastatic solid tumors known to have approved therapies using immune checkpoint inhibitors or anti-vascular endothelial growth factor agents
* Have exhausted (or refuse) all available standard of care therapy (e.g., including anti-PD1/programmed death ligand 1 [PDL1] if applicable) or for whom no standard therapy is available for their tumor type
* Patients with prior anti-PD1/PDL1 must have documentation of primary or secondary resistance to last prior anti-PD1/PDL1 therapy according to Immunotherapy Resistance Committee (SITC) (Kluger et al, 2020)
* Have at least 1 measurable lesion by RECIST 1.1 that has not been previously irradiated (for Part 2 only)
* Have recently obtained archival tumor tissue sample available, or undergo de novo tumor biopsy
* Eastern Cooperative Oncology Group (ECOG) PS 0-1
* Adequate hematologic, renal, and liver functions
* Dose Escalation (Part 1A and 1B): Any advanced or metastatic solid tumor fulfilling other relevant eligibility criteria.
* Dose Expansion (Part 2): Tumor specific cohorts (NSCLC, RCC, melanoma, MSS CRC) must have received prior approved therapies (Part 2)

Exclusion Criteria:

* Other active malignancy
* Recent major surgery
* Systemic anticancer therapy and chemotherapy within protocol-defined washout period
* Known or suspected hypersensitivity to prior treatment with any vaccinia oncolytic, pox virus, or antiviral agents within the past 10 years
* Current or history of myocarditis or congestive heart failure (New York Heart Association [NYHA] III-IV); unstable angina; or serious uncontrolled arrhythmia or recent myocardial infarction
* Active or history of interstitial lung disease (ILD)/pneumonitis
* Patients requiring chronic systemic immunosuppressants
* History of severe immune mediated side effect that was considered related to prior immune modulatory therapy and requiring immunosuppressive therapy
* Known symptomatic brain metastases requiring steroids
* History of or ongoing severe inflammatory skin conditions or severe eczema having required medical treatment
* Any prior or planned organ transplant
* Presence of any open, active wound requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Columbia University Medical Center, New York, New York
  - CUMC Research Pharmacy, New York, New York

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4651001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was planned to be conducted in 2 parts: Part 1 dose escalation for PF-07263689 monotherapy (Part 1A) and combination with sasanlimab (Part 1B) and Part 2 dose expansion for the combination therapy. The study was terminated during Part 1A due to sponsor's business decision; hence, Part 1B and Part 2 were not conducted and no participants were enrolled in Part 1B and 2.
Pre-assignment Details: A total of 13 participants were enrolled in Part 1A of the study.
Groups:
- Part 1A PF-07263689 2*10^8 PFU: Participants with any advanced or metastatic solid tumor indications with approved therapies using immune checkpoint inhibitors or anti-vascular endothelial growth factor agents were administered PF-07263689 at a dose 2*10^8 plaque forming unit (PFU) once weekly for 4 weeks as an intravenous (IV) push. Participants were followed up for up to 90 days post-last dose of study treatment. Participants were followed up for survival until death, withdrawal of consent, or end of the study.
- Part 1A PF-07263689 6*10^8 PFU: Participants with any advanced or metastatic solid tumor indications with approved therapies using immune checkpoint inhibitors or anti-vascular endothelial growth factor agents were administered PF-07263689 at a dose 6*10^8 PFU once weekly for 4 weeks as an IV push. Participants were followed up for up to 90 days post-last dose of study treatment. Participants were followed up for survival until death, withdrawal of consent, or end of the study.
- Part 1A PF-07263689 20*10^8PFU: Participants with any advanced or metastatic solid tumor indications with approved therapies using immune checkpoint inhibitors or anti-vascular endothelial growth factor agents were administered PF-07263689 at a dose 20*10^8 PFU once weekly for 4 weeks as an IV push. Participants were followed up for up to 90 days post-last dose of study treatment. Participants were followed up for survival until death, withdrawal of consent, or end of the study.
- Part 1B: PF-07263689 + Sasanlimab: Participants were planned to receive escalating doses of PF-07263689 in combination with sasanlimab.
- Part 2: PF-07263689 + Sasanlimab: Participants were planned to receive PF-07263689 in combination with sasanlimab at the preliminary combination recommended Phase 2 dose from Part 1B.
Period: Treatment Phase
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU | Part 1B: PF-07263689 + Sasanlimab | Part 2: PF-07263689 + Sasanlimab
Started | 3 | 4 | 6 | 0 | 0
Completed | 3 | 2 | 2 | 0 | 0
Not Completed | 0 | 2 | 4 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0
Not completed — Global deterioration of health status | 0 | 1 | 0 | 0 | 0
Period: Follow up
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU | Part 1B: PF-07263689 + Sasanlimab | Part 2: PF-07263689 + Sasanlimab
Started | 3 | 3 (Eligible participants attended follow-up visit 28 to 90 days after discontinuation of study treatment.) | 4 (Eligible participants attended follow-up visit 28 to 90 days after discontinuation of study treatment.) | 0 | 0
Completed | 1 | 3 | 0 | 0 | 0
Not Completed | 2 | 0 | 4 | 0 | 0
Not completed — Other | 2 | 0 | 2 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 2 | 0 | 0
Period: Long-term Follow-up
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU | Part 1B: PF-07263689 + Sasanlimab | Part 2: PF-07263689 + Sasanlimab
Started | 2 (Eligible participants entered long term follow-up for survival.) | 3 | 2 (Eligible participants entered long term follow-up for survival.) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 2 | 0 | 0
Not completed — Study terminated by sponsor | 2 | 2 | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who received at least one dose of study intervention. Data was not collected for Part 1B and Part 2 as no participants were enrolled due to early termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU | Part 1B: PF-07263689 + Sasanlimab | Part 2: PF-07263689 + Sasanlimab | Total
Number analyzed (Participants) | 3 | 4 | 6 | 0 | 0 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (6.43) | 61.0 (6.78) | 47.3 (9.40) |  |  | 53.6 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 0 | 0 | 6
  Male | 2 | 3 | 2 | 0 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 3 | 0 | 0 | 8
  Not Hispanic or Latino | 2 | 0 | 3 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 2
  White | 1 | 3 | 5 | 0 | 0 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs=occurrence of any of following adverse events (AEs) attributable to PF-07263689 in first cycle (cycle=28 days): Hematologic: grade(G)4 neutropenia lasting >5 days; febrile neutropenia; G3 neutropenia with infection, thrombocytopenia with bleeding; G4 thrombocytopenia. Non-hematologic: any treatment-related G>=3 toxicity; clinical events consistent with Hy's law; any G3 cytokine release syndrome (CRS) not improving to G<=2 within 72 hours despite medical management; any G4 CRC; G>=3 toxicity of any duration affecting vital organs; G4 vaccinia infection lasting >=6 days; G>=3 toxicities persisting for >3 days despite medical therapy (e.g. nausea, vomiting, diarrhea, fatigue); G >=3 rash not resolving to G<2 within 21 days with supportive measures; G>=3 lab abnormalities not controlled to G <=2 with or without appropriate medical management within 3 days; treatment-related AE inducing a delay by 2 weeks in receiving next scheduled dose; clinically important or persistent toxicities.
Time Frame: Up to 28 days
Population: DLT evaluable set included participants who received 3 of the 4 doses of PF-07263689 and had completed the scheduled safety assessments during the DLT observation period or had experienced a DLT. Data is not reported for Part 1b as no participants were enrolled and data was not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 3 | 4
Participants | 0 | 0 | 0

2. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Treatment Related Treatment Emergent Adverse Events and Treatment Related Serious Adverse Events
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was defined as any untoward medical occurrence that at any dose met 1 or more of the following criteria: resulted in death, was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic; an important medical event; required inpatient hospitalization or prolongation of existing hospitalization. TEAE was defined as any adverse event that occurred during the on-treatment period, on or after the first dose of study treatment. Relatedness was based on investigator's assessment.
Time Frame: From first dose of study treatment until 90 days after last dose of study treatment or before start of new anti-cancer therapy (up to maximum of 10.45 months)
Population: Safety analysis set included all enrolled participants who received at least one dose of study treatment. Data is not reported for Part 1b as no participants were enrolled and data was not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Participants
  TEAEs | 3 | 4 | 6
  SAEs | 0 | 1 | 2
  Treatment related TEAEs | 2 | 3 | 6
  Treatment related SAEs | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events Based on Maximum Common Terminology Criteria for Adverse Events (CTCAE) Version 5 Grade
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAE was defined as any AE that occurred during the on-treatment period, on or after the first dose of study treatment. AEs were graded using CTCAE version 5 where, grade 1=mild AE; grade 2=moderate AE; grade 3=severe AE; grade 4= life-threatening; urgent intervention indicated; and grade 5= death related to AE.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Participants
  Grade 1 | 3 | 2 | 1
  Grade 2 | 0 | 0 | 1
  Grade 3 | 0 | 2 | 4
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

4. Primary Outcome: Part 1: Number of Participants With Hematology Abnormalities by Maximum On-Treatment CTCAE Grade
Description: Hematology abnormalities were graded using CTCAE version 5 where, grade 0=non-missing lab value outside the grading range for the corresponding lab parameter; grade 1=mild; grade 2=moderate; grade 3=severe; grade 4= life-threatening. Only those categories with non-zero values for any of the arms have been reported.
Time Frame: From first dose of study treatment until 1 month follow-up (28+/-7) days after last dose of study treatment (up to 24 days of treatment exposure)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Participants
  Activated PTT prolonged: Grade 0 | 2 | 2 | 3
  Activated PTT prolonged: Grade 1 | 1 | 1 | 3
  Activated PTT prolonged: Grade 2 | 0 | 1 | 0
  Anemia: Grade 0 | 1 | 1 | 0
  Anemia: Grade 1 | 1 | 1 | 4
  Anemia: Grade 2 | 1 | 0 | 1
  Anemia: Grade 3 | 0 | 2 | 1
  Hemoglobin increased: Grade 0 | 3 | 4 | 6
  INR increased: Grade 0 | 3 | 3 | 5
  INR increased: Grade 1 | 0 | 1 | 1
  Leukocytosis: Grade 0 | 3 | 4 | 6
  Lymphocyte count decreased: Grade 0 | 1 | 0 | 0
  Lymphocyte count decreased: Grade 2 | 0 | 4 | 2
  Lymphocyte count decreased: Grade 3 | 2 | 0 | 4
  Lymphocyte count increased: Grade 0 | 3 | 4 | 6
  Neutrophil count decreased: Grade 0 | 1 | 4 | 5
  Neutrophil count decreased: Grade 1 | 2 | 0 | 0
  Neutrophil count decreased: Grade 2 | 0 | 0 | 1
  Platelet count decreased: Grade 0 | 2 | 2 | 4
  Platelet count decreased: Grade 1 | 1 | 2 | 2
  White blood cell decreased: Grade 0 | 3 | 4 | 3
  White blood cell decreased: Grade 1 | 0 | 0 | 2
  White blood cell decreased: Grade 2 | 0 | 0 | 1

5. Primary Outcome: Part 1: Number of Participants With Clinical Chemistry Abnormalities by Maximum On-Treatment CTCAE Grade
Description: Clinical chemistry abnormalities were graded using CTCAE version 5 where, grade 0=non-missing lab value outside the grading range for the corresponding lab parameter; grade 1=mild; grade 2=moderate; grade 3=severe; grade 4= life-threatening. Only those categories with non-zero values for any of the arms have been reported.
Time Frame: as for outcome 4
Population: Safety analysis set included all enrolled participants who received at least one dose of study treatment. Data is not reported for Part 1b as no participants were enrolled and data was not collected. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Participants
  Alanine aminotransferase increased: Grade 0 | 3 | 3 | 4
  Alanine aminotransferase increased: Grade 1 | 0 | 1 | 2
  Alkaline phosphatase increased: Grade 0 | 2 | 3 | 4
  Alkaline phosphatase increased: Grade 1 | 1 | 1 | 2
  Aspartate aminotransferase increased: Grade 0 | 3 | 3 | 5
  Aspartate aminotransferase increased: Grade 1 | 0 | 1 | 1
  Blood bilirubin increased: Grade 0 | 3 | 3 | 4
  Blood bilirubin increased: Grade 1 | 0 | 1 | 2
  Creatinine phosphokinase increased: Grade 0: number analyzed (Participants) | 2 | 4 | 6
  Creatinine phosphokinase increased: Grade 0 | 2 | 4 | 5
  Creatinine phosphokinase increased: Grade 1: number analyzed (Participants) | 2 | 4 | 6
  Creatinine phosphokinase increased: Grade 1 | 0 | 0 | 1
  Cardiac Troponin I Increased: Grade 0: number analyzed (Participants) | 3 | 3 | 5
  Cardiac Troponin I Increased: Grade 0 | 3 | 3 | 5
  Cardiac Troponin T Increased: Grade 0: number analyzed (Participants) | 0 | 1 | 1
  Cardiac Troponin T Increased: Grade 0 |  | 1 | 0
  Cardiac Troponin T Increased: Grade 1: number analyzed (Participants) | 0 | 1 | 1
  Cardiac Troponin T Increased: Grade 1 |  | 0 | 1
  Creatinine increased: Grade 0 | 2 | 4 | 4
  Creatinine increased: Grade 2 | 1 | 0 | 2
  Hypercalcemia: Grade 0 | 3 | 4 | 6
  Hyperkalemia: Grade 0 | 3 | 4 | 5
  Hyperkalemia: Grade 2 | 0 | 0 | 1
  Hypermagnesemia: Grade 0 | 3 | 4 | 6
  Hypernatremia: Grade 0 | 3 | 4 | 6
  Hypoalbuminemia: Grade 0 | 2 | 1 | 2
  Hypoalbuminemia: Grade 1 | 1 | 3 | 2
  Hypoalbuminemia: Grade 2 | 0 | 0 | 2
  Hypocalcemia: Grade 0 | 3 | 4 | 5
  Hypocalcemia: Grade 1 | 0 | 0 | 1
  Hypoglycemia: Grade 0 | 2 | 3 | 3
  Hypoglycemia: Grade 1 | 1 | 1 | 2
  Hypoglycemia: Grade 3 | 0 | 0 | 1
  Hypokalemia: Grade 0 | 2 | 2 | 4
  Hypokalemia: Grade 2 | 1 | 2 | 2
  Hypomagnesemia: Grade 0 | 2 | 3 | 4
  Hypomagnesemia: Grade 1 | 1 | 1 | 2
  Hyponatremia: Grade 0 | 1 | 0 | 1
  Hyponatremia: Grade 1 | 2 | 4 | 4
  Hyponatremia: Grade 3 | 0 | 0 | 1

6. Primary Outcome: Part 2: Number of Participants With Treatment Emergent Adverse Events, Serious Adverse Events, Treatment Related Treatment Emergent Adverse Events and Treatment Related Serious Adverse Events
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was defined as any untoward medical occurrence that at any dose met 1 or more of the following criteria: resulted in death, was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic; an important medical event; required inpatient hospitalization or prolongation of existing hospitalization. TEAE was defined as any adverse event that occurred during the on-treatment period, on or after the first dose of study treatment. Relatedness was planned to be assessed by investigator.
Time Frame: From first dose of study treatment until 90 days after last dose of study treatment or before start of new anti-cancer therapy (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

7. Primary Outcome: Part 2: Number of Participants With Treatment Emergent Adverse Events Based on Maximum CTCAE Version 5 Grade
Description: AEs were planned to be graded using CTCAE version 5 where, grade 1=mild AE; grade 2=moderate AE; grade 3=severe AE; grade 4= life-threatening; urgent intervention indicated; and grade 5= death related to AE.
Time Frame: as for outcome 6
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

8. Primary Outcome: Part 2: Number of Participants With Laboratory Abnormalities by Maximum On-Treatment CTCAE Grade
Description: Hematology and clinical chemistry parameters were planned to be assessed.
Time Frame: From first dose of study treatment until 35 days after last dose of study treatment or before start of new anti-cancer therapy (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

9. Primary Outcome: Part 2: Objective Response Rate
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) and was determined using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 millimeter [mm] short axis), PR: at least 30 percent (%) decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions.
Time Frame: From first dose of study treatment until CR or PR (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

10. Secondary Outcome: Part 1: Objective Response Rate
Description: ORR was defined as the percentage of participants with a best overall response of CR or PR and was determined using RECIST version 1.1. CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 mm short axis), PR: at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. 95% confidence interval (CI) was based on Clopper-Pearson method.
Time Frame: From first dose of study treatment until CR or PR (up to maximum follow-up of 10.45 months)
Population: Response evaluable set included all participants who received at least one dose of study treatment and had baseline disease assessment [or measurable disease at baseline, if applicable] and at least one post-baseline disease assessment. Data is not reported for Part 1b as no participants were enrolled and data was not collected.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 3 | 4
Percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2]

11. Secondary Outcome: Part 1: Duration of Response
Description: Duration of response was defined as the time from first documentation of CR or PR to date of first documentation of progressive disease (PD) or death due to any cause. CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non- pathological in size (<10 mm short axis), PR: at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. PD: 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm and unequivocal progression of pre-existing lesions.
Time Frame: From first documentation of CR or PR to date of first documentation of PD or death due to any cause (up to maximum follow-up of 10.45 months)
Population: Response evaluable set included all participants who received at least one dose of study treatment and had baseline disease assessment [or measurable disease at baseline, if applicable] and at least one post-baseline disease assessment. Only participants with CR or PR were analyzed. Data is not reported for Part 1b as no participants were enrolled and data was not collected.
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Part 1: Progression Free Survival
Description: Progression free survival was defined as time from start date of treatment to the date of first documentation of PD or death due to any cause. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm and unequivocal progression of pre-existing lesions. 95% CI was based on Brookmeyer and Crowley method.
Time Frame: From start date of treatment to the date of first documentation of PD or death due to any cause (up to maximum follow-up of 10.45 months)
Population: Full analysis set included all enrolled participants. Data is not reported for Part 1b as no participants were enrolled and data was not collected.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Months | 1.4 [1.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 1.5 [1.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 1.4 [1.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.

13. Secondary Outcome: Part 1: Time to Progression
Description: Time to progression was defined as the time from start date of treatment to the date of the first documentation of PD. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm and unequivocal progression of pre-existing lesions. 95% CI was based on Brookmeyer and Crowley method.
Time Frame: From start date of treatment to the date of first documentation of PD (up to maximum follow-up of 10.45 months)
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Months | 1.4 [1.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 1.5 [1.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 1.4 [1.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.

14. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) of PF-07263689 in Blood
Time Frame: Day 1 (pre-dose, 0.5, 1, 4, 8 hours post-dose), Day 2, Day 3, Day 4, Day 8 (pre-dose, 0.5, 1, 4, 8 hours post-dose), Day 9, Day 10, Day 15 and 22 (pre-dose and 4 hours post-dose)
Population: Blood viral load Kinetics Analysis Set included all enrolled participants treated who did not have protocol deviations influencing viral load kinetics assessment, and had sufficient information to estimate at least 1 of the parameters of interest. Data is not reported for Part 1b as no participants were enrolled and data was not collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per milliliter
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Copies per milliliter | NA (NA) — Cmax could not be calculated as the values were below limit of quantification. | NA (NA) — Cmax could not be calculated as the values were below limit of quantification. | NA (NA) — Cmax could not be calculated as the values were below limit of quantification.

15. Secondary Outcome: Part 1: Time to Maximum Concentration (Tmax) of PF-07263689 in Blood
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Hours | NA [NA to NA] — Tmax could not be calculated as the values were below limit of quantification. | NA [NA to NA] — Tmax could not be calculated as the values were below limit of quantification. | NA [NA to NA] — Tmax could not be calculated as the values were below limit of quantification.

16. Secondary Outcome: Part 1: Area Under the Concentration-Time Curve From Time 0 to Time of Last Measurable Concentration of PF-07263689 in Blood
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*copies per milliliter
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Hours*copies per milliliter | NA (NA) — AUC(0 to t) could not be calculated as the values were below limit of quantification. | NA (NA) — AUC(0 to t) could not be calculated as the values were below limit of quantification. | NA (NA) — AUC(0 to t) could not be calculated as the values were below limit of quantification.

17. Secondary Outcome: Part 1b: Trough Concentration of Sasanlimab
Time Frame: pre-dose on Day 1, 8, 15 and 22
Population: Data was not collected as no participants were enrolled in Part 1b of the study due to study termination.
Arm/Group | Part 1B: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

18. Secondary Outcome: Part 1: Viral Titers in Saliva, Urine and Skin Swabs During 30, 45 and 60 Days After the Last PF-07263689 Dose
Description: Viral titers in each matrix (saliva, urine and skin swabs [30 days post last dose only]) at 30, 45 and 60 days after last dose of study treatment is reported in this outcome measure.
Time Frame: At 30, 45 and 60 days post last dose of study treatment (up to 24 days of treatment exposure)
Population: Vector Shedding Analysis Set included all enrolled participants who were treated and had at least 1 analyte concentration above the lower limit of quantitation. Data is not reported for Part 1b as no participants were enrolled and data was not collected. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and contributed data to the table and 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Copies per milliliter
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Copies per milliliter
  Saliva; 30 days post last dose: number analyzed (Participants) | 3 | 1 | 0
  Saliva; 30 days post last dose | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification. |
  Saliva; 45 days post last dose: number analyzed (Participants) | 3 | 3 | 1
  Saliva; 45 days post last dose | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification.
  Saliva; 60 days post last dose: number analyzed (Participants) | 3 | 3 | 0
  Saliva; 60 days post last dose | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification. |
  Skin swab; 30 days post last dose: number analyzed (Participants) | 3 | 1 | 0
  Skin swab; 30 days post last dose | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification. |
  Urine; 30 days post last dose: number analyzed (Participants) | 3 | 1 | 0
  Urine; 30 days post last dose | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification. |
  Urine; 45 days post last dose: number analyzed (Participants) | 3 | 3 | 1
  Urine; 45 days post last dose | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification.
  Urine; 60 days post last dose: number analyzed (Participants) | 3 | 3 | 0
  Urine; 60 days post last dose | NA (NA) — Data could not be calculated as the values were below the limit of quantification. | NA (NA) — Data could not be calculated as the values were below the limit of quantification. |

19. Secondary Outcome: Part 1: Percentage of Participants With Positive Neutralizing Antibodies Against PF-07263689 and Sasanlimab
Description: A participant was considered NAb positive if (1) baseline titer was missing or negative and participant had >= 1 post-treatment positive titer (treatment-induced) or (2) positive titer at baseline and had a ratio of >= 4 in titer (dilution) to baseline in >= 1 post-treatment sample (treatment-boosted). Percentage of participants with positive neutralizing antibodies against PF-07263689 is presented in this outcome measure. Data was not collected for sasanlimab as no participants were enrolled in Part 1b of the study.
Time Frame: From Baseline (pre-dose) on Day 1 up to Day 22
Population: Immunogenicity analysis set included all enrolled participants who received at least one dose of study treatment and had at least one sample tested for ADA. Data is not reported for Part 1b as no participants were enrolled and data was not collected.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Percentage of participants | 66.7 | 50.0 | 100.0

20. Secondary Outcome: Part 1: Percentage of Participants With Positive Anti-interleukin 2 Antibodies
Description: A participant was considered anti-drug antibody (ADA) positive if (1) baseline titer was missing or negative and participant had >= 1 post-treatment positive titer (treatment-induced) or (2) positive titer at baseline and had a ratio of >= 4 in titer (dilution) to baseline in >= 1 post-treatment sample (treatment-boosted). Percentage of participants with positive anti-interleukin 2 antibodies against PF-07263689 is presented in this outcome measure.
Time Frame: From Baseline (pre-dose) on Day 1 up to Day 22
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU
Number analyzed (Participants) | 3 | 4 | 6
Percentage of participants | 0.0 | 25.0 | 0.0

21. Secondary Outcome: Part 2: Maximum Observed Concentration (Cmax) of PF-7263689 in Blood
Time Frame: as for outcome 14
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

22. Secondary Outcome: Part 2: Time to Maximum Concentration (Tmax) of PF-07263689 in Blood
Time Frame: as for outcome 14
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

23. Secondary Outcome: Part 2: Area Under the Concentration-Time Curve From Time 0 to Time of Last Measurable Concentration of PF-07263689 in Blood
Time Frame: as for outcome 14
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

24. Secondary Outcome: Part 2: Trough Concentration of Sasanlimab
Time Frame: Pre-dose on Day 1, 8, 15 and 22
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

25. Secondary Outcome: Part 2: Viral Titers in Saliva, Urine and Skin Swabs During 30, 45 and 60 Days After the Last PF-07263689 Dose
Time Frame: 30, 45 and 60 days after the last PF-07263689 dose
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

26. Secondary Outcome: Part 2: Percentage of Participants With Positive Anti-drug Antibodies Against PF-07263689 and Sasanlimab
Time Frame: From first dose of study treatment until 60 days after last dose of study treatment (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

27. Secondary Outcome: Part 2: Titer for Anti-PF-07263689 Antibody
Time Frame: From first dose of study treatment until 60 days after last dose of study treatment (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

28. Secondary Outcome: Part 2: Percentage of Participants With Positive Anti-interleukin 2 Antibodies
Time Frame: From first dose of study treatment until 60 days after last dose of study treatment (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

29. Secondary Outcome: Part 2: Titer for Anti-IL2 Antibodies
Time Frame: From first dose of study treatment until 60 days after last dose of study treatment (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

30. Secondary Outcome: Part 2: Disease Control Rate
Description: Disease control rate was the percentage of participants with CR, PR or stable disease (SD), as defined by RECIST 1.1. CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 mm short axis), PR: at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. SD: Does not qualify for CR, PR, or progression. All target lesions assessed.
Time Frame: From start of study treatment until CR, PR or SD (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

31. Secondary Outcome: Part 2: Duration of Response
Description: as for outcome 11
Time Frame: From first documentation of CR or PR to date of first documentation of PD or death due to any cause (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

32. Secondary Outcome: Part 2: Progression Free Survival
Description: Progression free survival was defined as time from start date of treatment to the date of first documentation of PD or death due to any cause. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm and unequivocal progression of pre-existing lesions.
Time Frame: From start date of treatment to the date of first documentation of PD or death due to any cause (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

33. Secondary Outcome: Part 2: Time to Progression
Description: Time to progression was defined as the time from start date of treatment to the date of the first documentation of PD. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm and unequivocal progression of pre-existing lesions.
Time Frame: From start date of treatment to the date of first documentation of PD (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

34. Secondary Outcome: Part 2: Overall Survival
Description: Overall survival was defined as the duration from the start of study treatment to the date of death from any cause.
Time Frame: From start of study treatment to the date of death from any cause (up to 2 years)
Population: Data was not collected as no participants were enrolled in Part 2 of the study due to study termination.
Arm/Group | Part 2: PF-07263689 + Sasanlimab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: From first dose of study treatment until death, withdrawal of consent, or end of the study (up to maximum follow-up of 10.45 months); SAEs and non-SAEs: From first dose of study treatment until 90 days after last dose of study treatment or before start of new anti-cancer therapy (up to maximum of 10.45 months).
Description: Same event may appear as both non-SAE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Adverse event reported only for Part 1a. Since there was no enrolment for Part 1b and 2, no safety data collected and reported.
Arm/Group | Part 1A PF-07263689 2*10^8 PFU | Part 1A PF-07263689 6*10^8 PFU | Part 1A PF-07263689 20*10^8PFU | Part 1B: PF-07263689 + Sasanlimab | Part 2: PF-07263689 + Sasanlimab
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 0/6 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 2/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A PF-07263689 2*10^8 PFU (N=3) | Part 1A PF-07263689 6*10^8 PFU (N=4) | Part 1A PF-07263689 20*10^8PFU (N=6) | Part 1B: PF-07263689 + Sasanlimab (N=0) | Part 2: PF-07263689 + Sasanlimab (N=0)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A PF-07263689 2*10^8 PFU (N=3) | Part 1A PF-07263689 6*10^8 PFU (N=4) | Part 1A PF-07263689 20*10^8PFU (N=6) | Part 1B: PF-07263689 + Sasanlimab (N=0) | Part 2: PF-07263689 + Sasanlimab (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 5 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 3 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 1 | 0 | 0
Induration (General disorders) | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 5 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 2 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 5 | 0 | 0
Slow speech (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 0 | 0

LIMITATIONS AND CAVEATS:
Data was not collected for Part 1B and Part 2 as no participants were enrolled due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05061537/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT05061537/SAP_001.pdf